CLINICAL TRIAL: NCT00052585
Title: A Phase II Trial Of IRESSA (NSC 715055, IND 61187) In Combination With 5-FU/LV/ CPT-11 In Patients With Advanced Or Recurrent Colorectal Cancer
Brief Title: Gefitinib and Combination Chemotherapy in Treating Patients With Advanced or Recurrent Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02505; UPCC #06202; CDR0000258548 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Gefitinib; Leucovorin; Fluorouracil

ARMS (1):
- Treatment (irinotecan, gefitinib, leucovorin, fluorouracil) (Experimental): Patients receive oral gefitinib daily beginning on day 1, irinotecan IV over 90 minutes on days 1 and 15, and leucovorin calcium IV over 2 hours and fluorouracil IV over 3-5 seconds followed by a 22-hour infusion on days 1, 2, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: gefitinib; Drug: leucovorin calcium; Drug: fluorouracil

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
Phase II trial to study the effectiveness of combining gefitinib with fluorouracil, leucovorin, and irinotecan in treating patients who have advanced or recurrent colorectal cancer. Biological therapies such as gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining gefitinib with fluorouracil, leucovorin, and irinotecan may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety of gefitinib, fluorouracil, leucovorin calcium, and irinotecan in patients with advanced or recurrent colorectal cancer.

II. Determine the major side effects of this regimen in these patients. III. Determine the response rate, progression-free survival, and overall survival of patients treated with this regimen.

IV. Correlate response and other measures of outcome with epidermal growth factor receptor expression and the expression of genes that impact upon pathways of fluoropyrimidine cytotoxicity in patients treated with this regimen.

OUTLINE: This is a non-randomized, open-label, multi-center study.

Patients receive oral gefitinib daily beginning on day 1, irinotecan IV over 90 minutes on days 1 and 15, and leucovorin calcium IV over 2 hours and fluorouracil IV over 3-5 seconds followed by a 22-hour infusion on days 1, 2, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced (stage IV) or recurrent adenocarcinoma of the colon or rectum
* Must have available tissue for immunohistochemical analysis
* At least one unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Tumor marker (carcinoembryonic antigen) elevation alone is insufficient for study entry
* No known brain metastases
* Performance status - ECOG 0-2
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST less than 2 times ULN (5 times ULN if liver involvement of tumor)
* Creatinine no greater than 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other severe or uncontrolled concurrent illness that would adversely impact the safety or efficacy of study therapy
* No ongoing or active infection
* No other prior malignancy unless curatively treated and no evidence of recurrence
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gefitinib
* No psychiatric illness or social situation that would preclude study compliance
* No prior chemotherapy for advanced disease
* More than 4 weeks since other prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 4 weeks since prior radiotherapy and recovered
* At least 6 months since prior adjuvant therapy
* No prior epidermal growth factor receptor inhibitor
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent phenytoin, carbamazepine, barbiturates, rifampin, rifapentine, oxacarbazepine, modafinil, griseofulvin, or Hypericum perforatum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-10; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Grade 3 or 4 toxicity, graded using the NCI CTC version 2.0 | Up to 2 years
Response rate | Up to 2 years
  95% confidence interval will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States